CLINICAL TRIAL: NCT00464412
Title: The Effect of a Short Educational Program on Young Women's Knowledge and Beliefs About Osteoporosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Valdosta State University (Other)
Collaborators: Roanoke College (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 1-Kasper
Record Dates: First submitted 2007-04-19; First posted 2007-04-23 (Estimated); Last update posted 2007-05-09 (Estimated); Status verified 2007-05

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; Knowledge; Beliefs; Education; Women
MeSH Terms: conditions — Osteoporosis | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Education

SUMMARY:
The purpose of the study is to determine the effect of a short educational program on young women's knowledge and beliefs about osteoporosis. They hypothesis is that following the intervention women who receive the educational program will have greater knowledge and beliefs about osteoporosis.

DETAILED DESCRIPTION:
Objective. To determine the effect of a short osteoporosis educational program on young women's knowledge and beliefs about osteoporosis. Methods. Ten college physical activity classes enrolling 133 predominantly Caucasian women (age range 18 to 21 years) were randomized to an osteoporosis educational program or control. Knowledge and beliefs about osteoporosis were assessed at baseline and at one week and three weeks following the intervention using the Multiple Osteoporosis Prevention Survey. Knowledge was defined as the ability to identify correctly osteoporosis risk factors. Beliefs were measured with the use of a five point Likert type scale. The educational program was comprised of a lecture and printed materials developed by the National Osteoporosis Foundation. Chi-square and analysis of variance evaluated for between group differences. Alpha was set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Women enrolled in a mid-atlantic college physical activity course

Exclusion Criteria:

* Unable to partake in three survey's and one educational lesson

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2006-01; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Osteoporosis Knowledge | 7 days and 21 days post educational intervention
Osteoporosis Beliefs | 7 days and 21 days post educational intervention

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Kasper, EdD, Principal Investigator — Valdosta State University